CLINICAL TRIAL: NCT05119738
Title: Immune Response to Third Dose of SARS-CoV-2 Vaccine in a Cohort of Cancer Patients on Active Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 210410004
Record Dates: First submitted 2021-11-10; First posted 2021-11-15 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2021-10

CONDITIONS: Sars-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; sinovac COVID-19 vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Three doses of BNT162b2.: Cancer patients on active cytotoxic treatment who received three doses of BNT162b2.
  Interventions: Biological: Three doses of BNT162b2 (observational)
- Two doses of Coronavac and one of BNT162b2.: Cancer patients on active cytotoxic treatment who received two doses of Coronavac and one dose of BNT162b2.
  Interventions: Biological: Two doses of Coronavac and one dose BNT162b2 (observational)

INTERVENTIONS:
Biological: Three doses of BNT162b2 (observational) — BNT162b2 (COVID 19 mRNA vaccine)
  Groups: Three doses of BNT162b2.
Biological: Two doses of Coronavac and one dose BNT162b2 (observational) — BNT162b2 (COVID 19 mRNA vaccine) Coronavac (COVID 19 inactive vaccine)
  Groups: Two doses of Coronavac and one of BNT162b2.

SUMMARY:
The Coronavirus Disease 2019 (COVID-19) pandemic has claimed over 5 million lives globally. Fortunately, a substantial and growing number of SARS-CoV-2 vaccines with very high efficacy have been developed, manufactured, and rapidly approved. Novel mRNA vaccines such as the BNT162b2 (Pfizer-BioNTech) and mRNA-1273 (Moderna) have reported a stunning >94% efficacy against COVID-19. However, global access has not been equitable, with many low- and middle-income countries having no vaccine access or access under emergency use mainly to traditional inactivated SARS-CoV2-2 vaccines such as BBIBP-CorV (Sinopharm Beijing), CoronaVac (Sinovac) and BBV152 (Bharat Biotech). Emerging studies have shown that lower concentrations of neutralizing antibodies (Nab) are attained after CoronaVac than after a mRNA-based vaccine in healthy individuals. This difference seems to be more pronounced in immunocompromised patients who are at higher risk of severe COVID-19 and death from COVID-19. As such several countries including United States, Israel and Chile have recommended a third vaccine dose for this vulnerable population.

In this observational study we will explore the humoral response to the BNT162b2 vaccine in patients who received two previous doses of the inactivated vaccine Coronavac or two doses of BNT162b2.

ELIGIBILITY:
Inclusion Criteria:

* Vaccination with two doses of Coronavac vaccine or BNT162b2 vaccine
* Eastern Cooperative Oncology group performance status < 3

Exclusion Criteria:

* Previous SARS-CoV-2 infection
* Vaccination with booster vaccine more than 12 weeks before informed consent
* Intravenous inmunoglobulin therapy 60 days before informed consent
* Any condition that could interfere with the paticipant´s participation during the study in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients receiving their care at the Red de Salud UC Christus in Santiago Chile will be invited
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of positive neutralizing antibodies 8 to 12 weeks after third dose BNT162b2 (booster vaccine). | 8 to12 weeks after third dose BNT162b2.

SECONDARY OUTCOMES:
Neutralizing geometric mean titers 8 to 12 weeks after third dose BNT162b2 (booster vaccine) | 8 to12 weeks after third dose BNT162b2.

CONTACTS AND LOCATIONS:
Locations (1):
- Red de Salud UC Christus, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No